CLINICAL TRIAL: NCT00466453
Title: Adapting Web-based Instruction to Learner Baseline Knowledge: A Randomized Controlled Trial
Brief Title: Adapting Web-based Instruction to Baseline Knowledge of Physicians-in-training
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 05-004123
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Medical Education; Medical Training; Internship and Residency

INTERVENTIONS:
Behavioral: knowledge-adaptive Web-based instruction

SUMMARY:
The purpose of this study is to compare an adaptive Web-based learning system to a non-adaptive system for teaching physicians-in-training about ambulatory medicine.

DETAILED DESCRIPTION:
Not all Web-based instruction is equally effective at facilitating learning. Adaptation to characteristics of individual learners may enhance Web-based learning by emulating a face-to-face teacher's response to a learner's needs. Learner baseline knowledge level is one variable to which Web-based instruction may adapt. We will enhance Web-based instructional modules used in the Internal Medicine resident continuity clinics so that they adapt to learner baseline knowledge. We will then compare the adaptive Web-based format to the standard format. We hypothesize that the adaptive format will have higher learning efficiency, and that achievement will be similar for the two groups. We also hypothesize that residents will prefer the adaptive format and find it to be more motivating than the standard format.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine residents (Mayo-Rochester campus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144
Dates: Start 2005-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Knowledge
Learning efficiency

SECONDARY OUTCOMES:
Format preference
Time to complete module
Motivation

CONTACTS AND LOCATIONS:
Overall Officials: David A. Cook, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Cook DA, Beckman TJ, Thomas KG, Thompson WG. Adapting web-based instruction to residents' knowledge improves learning efficiency: a randomized controlled trial. J Gen Intern Med. 2008 Jul;23(7):985-90. doi: 10.1007/s11606-008-0541-0. PMID 18612729